CLINICAL TRIAL: NCT03473249
Title: Clinical Effectiveness of Contrast-Enhanced Ultrasound in the Evaluation of Blunt Abdominal Trauma in Young Children
Brief Title: Effectiveness of Contrast-Enhanced Ultrasound
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-014183
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Injuries; Physical Abuse; Accidental Fall; Motor Vehicle Injury
MeSH Terms: conditions — Abdominal Injuries | interventions — contrast agent BR1; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Retrospective Review (No Intervention): Comparison of CT and CEUS results from retrospective chart review of children who have had a CEUS for trauma at the Children's Hospital of Philadelphia (CHOP).
- Prospective Observation (No Intervention): Prospective observation of comparison of CT and CEUS results among children who are undergoing a CEUS and abdominal CT as part of clinical care.
- Contrast-Enhanced Ultrasound using Lumason (Other): Prospective intervention using contrast enhanced ultrasound with IV contrast Lumason.
  Interventions: Drug: Contrast-Enhanced Ultrasound using Lumason

INTERVENTIONS:
Drug: Contrast-Enhanced Ultrasound using Lumason — Subjects will undergo a contrast enhanced ultrasound (CEUS) during which a standard greyscale abdominal ultrasound is performed first followed by injection of intravenous contrast with Lumason, and completion of contrast-enhanced ultrasound
  Other Names: SonoVue (25 mg under sulfur hexafluoride gas) / Lumason; Sulfur hexafluoride microbubbles for injection; US Patent No. 5,686,060
  Arms: Contrast-Enhanced Ultrasound using Lumason

SUMMARY:
The purpose of the study is to generate pilot data describing test characteristics of contrast enhanced ultrasound in young children with concern for abdominal trauma. The primary objective in this study is to determine the sensitivity and specificity of contrast-enhanced ultrasound (CEUS) compared to abdominal Computed Tomography (CT) in the detection of abdominal solid organ injury in young children < 8 years of age with concern for blunt abdominal trauma.

DETAILED DESCRIPTION:
Abdominal trauma in children can be deadly, but intra-abdominal injuries can be difficult to detect and often lack external signs of injury on physical exam. The current gold standard imaging study is Computed Tomography (CT) with IV contrast, which is associated with radiation exposure. Contrast-enhanced ultrasound is a radiation-free alternative to detect abdominal injuries and has been studied primarily in adults and some older children, but evidence to support its use in young children is needed.

This is a prospective study of children less than 8 years of age who are clinically stable and undergoing an abdominal CT with IV contrast as part of their clinical care due to concerns for abdominal trauma. Investigators will compare CEUS results with those obtained by CT. Investigators will additionally include retrospective data of children who underwent both abdominal CT and CEUS as part of clinical care.

ELIGIBILITY:
Inclusion Criteria for study CEUS

1. Males or females < 8 years of age at time of enrollment
2. Clinically stable (defined as not undergoing an emergent surgical procedure in the next hour)
3. Abdominal CT ordered or obtained
4. IV in place

Exclusion Criteria for study CEUS

1. Unable to obtain contrast-enhanced ultrasound within 72 hours after CT
2. History of allergic reaction to Lumason, sulfa-hexafluoride lipid microsphere components, or other ingredients in Lumason (polyethylene glycol 4000, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na) palmitic acid)
3. Known congenital or acquired heart disease

Alternative Inclusion and Exclusion Criteria for children who have undergone or are undergoing CEUS as part of clinical care

Inclusion criteria:

1. Males or females < 8 years of age at time of CEUS.
2. Clinical Team plans to perform CT or has performed CT as part of clinical care for abdominal trauma
3. Clinical Team plans to perform (or has performed) CEUS as part of clinical care
4. Date of CEUS after January 1, 2015

Exclusion Criteria: None

Ages: 0 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Contrast-Enhanced Ultrasound in detection of abdominal solid organ injury in young children <8 years of age | 2 years
  To determine the sensitivity of contrast-enhanced ultrasound (CEUS) compared with standard, abdominal Computer Tomography (CT) in the detection of abdominal solid organ injury in young children < 8 years of age with concern for blunt abdominal trauma.
Specificity of Contrast-Enhanced Ultrasound in detection of abdominal solid organ injury in young children <8 years of age | 2 years
  To determine the specificity of contrast-enhanced ultrasound (CEUS) compared with standard, abdominal Computer Tomography (CT) in the detection of abdominal solid organ injury in young children < 8 years of age with concern for blunt abdominal trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wood J, Rubin DM, Nance ML, Christian CW. Distinguishing inflicted versus accidental abdominal injuries in young children. J Trauma. 2005 Nov;59(5):1203-8. doi: 10.1097/01.ta.0000196437.07011.b1. PMID 16385300
- [Background] Lutz N, Nance ML, Kallan MJ, Arbogast KB, Durbin DR, Winston FK. Incidence and clinical significance of abdominal wall bruising in restrained children involved in motor vehicle crashes. J Pediatr Surg. 2004 Jun;39(6):972-5. doi: 10.1016/j.jpedsurg.2004.02.029. PMID 15185237
- [Background] Carter KW, Moulton SL. Pediatric abdominal injury patterns caused by "falls": A comparison between nonaccidental and accidental trauma. J Pediatr Surg. 2016 Feb;51(2):326-8. doi: 10.1016/j.jpedsurg.2015.10.056. Epub 2015 Oct 31. PMID 26850907
- [Background] Cooper A, Floyd T, Barlow B, Niemirska M, Ludwig S, Seidl T, O'Neill J, Templeton J, Ziegler M, Ross A, et al. Major blunt abdominal trauma due to child abuse. J Trauma. 1988 Oct;28(10):1483-7. doi: 10.1097/00005373-198810000-00015. PMID 3172310
- [Background] Lindberg D, Makoroff K, Harper N, Laskey A, Bechtel K, Deye K, Shapiro R; ULTRA Investigators. Utility of hepatic transaminases to recognize abuse in children. Pediatrics. 2009 Aug;124(2):509-16. doi: 10.1542/peds.2008-2348. Epub 2009 Jul 20. PMID 19620197
- [Background] Lindberg DM, Shapiro RA, Blood EA, Steiner RD, Berger RP; ExSTRA investigators. Utility of hepatic transaminases in children with concern for abuse. Pediatrics. 2013 Feb;131(2):268-75. doi: 10.1542/peds.2012-1952. Epub 2013 Jan 14. PMID 23319537
- [Background] Trout AT, Strouse PJ, Mohr BA, Khalatbari S, Myles JD. Abdominal and pelvic CT in cases of suspected abuse: can clinical and laboratory findings guide its use? Pediatr Radiol. 2011 Jan;41(1):92-8. doi: 10.1007/s00247-010-1847-8. Epub 2010 Oct 9. PMID 20936274
- [Background] Hennes HM, Smith DS, Schneider K, Hegenbarth MA, Duma MA, Jona JZ. Elevated liver transaminase levels in children with blunt abdominal trauma: a predictor of liver injury. Pediatrics. 1990 Jul;86(1):87-90. PMID 2359686
- [Background] Rothrock SG, Green SM, Morgan R. Abdominal trauma in infants and children: prompt identification and early management of serious and life-threatening injuries. Part I: injury patterns and initial assessment. Pediatr Emerg Care. 2000 Apr;16(2):106-15. doi: 10.1097/00006565-200004000-00012. PMID 10784214
- [Background] Goske MJ, Applegate KE, Bulas D, Butler PF, Callahan MJ, Coley BD, Don S, Frush DP, Hernanz-Schulman M, Kaste SC, Morrison G, Sidhu M, Strauss KJ, Treves ST; Alliance for Radiation Safety in Pediatric Imaging. Image Gently: progress and challenges in CT education and advocacy. Pediatr Radiol. 2011 Sep;41 Suppl 2:461-6. doi: 10.1007/s00247-011-2133-0. Epub 2011 Aug 17. PMID 21847723
- [Background] Laugesen NG, Nolsoe CP, Rosenberg J. Clinical Applications of Contrast-Enhanced Ultrasound in the Pediatric Work-Up of Focal Liver Lesions and Blunt Abdominal Trauma: A Systematic Review. Ultrasound Int Open. 2017 Feb;3(1):E2-E7. doi: 10.1055/s-0042-124502. PMID 28255580
- [Background] Miele V, Piccolo CL, Trinci M, Galluzzo M, Ianniello S, Brunese L. Diagnostic imaging of blunt abdominal trauma in pediatric patients. Radiol Med. 2016 May;121(5):409-30. doi: 10.1007/s11547-016-0637-2. Epub 2016 Apr 13. PMID 27075018
- [Background] Catalano O, Aiani L, Barozzi L, Bokor D, De Marchi A, Faletti C, Maggioni F, Montanari N, Orlandi PE, Siani A, Sidhu PS, Thompson PK, Valentino M, Ziosi A, Martegani A. CEUS in abdominal trauma: multi-center study. Abdom Imaging. 2009 Mar-Apr;34(2):225-34. doi: 10.1007/s00261-008-9452-0. PMID 18682877
- [Background] Clevert DA, Weckbach S, Minaifar N, Clevert DA, Stickel M, Reiser M. Contrast-enhanced ultrasound versus MS-CT in blunt abdominal trauma. Clin Hemorheol Microcirc. 2008;39(1-4):155-69. PMID 18503121
- [Background] Manetta R, Pistoia ML, Bultrini C, Stavroulis E, Di Cesare E, Masciocchi C. Ultrasound enhanced with sulphur-hexafluoride-filled microbubbles agent (SonoVue) in the follow-up of mild liver and spleen trauma. Radiol Med. 2009 Aug;114(5):771-9. doi: 10.1007/s11547-009-0406-6. Epub 2009 May 30. English, Italian. PMID 19484583
- [Background] Thorelius L. Emergency real-time contrast-enhanced ultrasonography for detection of solid organ injuries. Eur Radiol. 2007 Dec;17 Suppl 6:F107-11. doi: 10.1007/s10406-007-0235-4. PMID 18376464
- [Background] Valentino M, Serra C, Zironi G, De Luca C, Pavlica P, Barozzi L. Blunt abdominal trauma: emergency contrast-enhanced sonography for detection of solid organ injuries. AJR Am J Roentgenol. 2006 May;186(5):1361-7. doi: 10.2214/AJR.05.0027. PMID 16632732
- [Background] Piscaglia F, Bolondi L; Italian Society for Ultrasound in Medicine and Biology (SIUMB) Study Group on Ultrasound Contrast Agents. The safety of Sonovue in abdominal applications: retrospective analysis of 23188 investigations. Ultrasound Med Biol. 2006 Sep;32(9):1369-75. doi: 10.1016/j.ultrasmedbio.2006.05.031. PMID 16965977
- [Background] Oldenburg A, Hohmann J, Skrok J, Albrecht T. Imaging of paediatric splenic injury with contrast-enhanced ultrasonography. Pediatr Radiol. 2004 Apr;34(4):351-4. doi: 10.1007/s00247-003-1092-5. Epub 2003 Dec 2. PMID 14652701
- [Background] Valentino M, Serra C, Pavlica P, Labate AM, Lima M, Baroncini S, Barozzi L. Blunt abdominal trauma: diagnostic performance of contrast-enhanced US in children--initial experience. Radiology. 2008 Mar;246(3):903-9. doi: 10.1148/radiol.2463070652. Epub 2008 Jan 14. PMID 18195385
- [Background] Menichini G, Sessa B, Trinci M, Galluzzo M, Miele V. Accuracy of contrast-enhanced ultrasound (CEUS) in the identification and characterization of traumatic solid organ lesions in children: a retrospective comparison with baseline US and CE-MDCT. Radiol Med. 2015 Nov;120(11):989-1001. doi: 10.1007/s11547-015-0535-z. Epub 2015 Mar 31. PMID 25822953
- [Background] Riccabona M. Application of a second-generation US contrast agent in infants and children--a European questionnaire-based survey. Pediatr Radiol. 2012 Dec;42(12):1471-80. doi: 10.1007/s00247-012-2472-5. Epub 2012 Oct 3. PMID 23052725
- [Background] Piskunowicz M, Kosiak W, Batko T, Piankowski A, Polczynska K, Adamkiewicz-Drozynska E. Safety of intravenous application of second-generation ultrasound contrast agent in children: prospective analysis. Ultrasound Med Biol. 2015 Apr;41(4):1095-9. doi: 10.1016/j.ultrasmedbio.2014.11.003. Epub 2015 Feb 18. PMID 25701526
- [Background] Yusuf GT, Sellars ME, Deganello A, Cosgrove DO, Sidhu PS. Retrospective Analysis of the Safety and Cost Implications of Pediatric Contrast-Enhanced Ultrasound at a Single Center. AJR Am J Roentgenol. 2017 Feb;208(2):446-452. doi: 10.2214/AJR.16.16700. Epub 2016 Dec 13. PMID 27959665
- [Background] Jacob J, Deganello A, Sellars ME, Hadzic N, Sidhu PS. Contrast enhanced ultrasound (CEUS) characterization of grey-scale sonographic indeterminate focal liver lesions in pediatric practice. Ultraschall Med. 2013 Dec;34(6):529-40. doi: 10.1055/s-0033-1355785. Epub 2013 Oct 16. PMID 24132647
- [Background] Bonini G, Pezzotta G, Morzenti C, Agazzi R, Nani R. Contrast-enhanced ultrasound with SonoVue in the evaluation of postoperative complications in pediatric liver transplant recipients. J Ultrasound. 2007 Jun;10(2):99-106. doi: 10.1016/j.jus.2007.02.008. Epub 2007 Jun 13. PMID 23396596
- [Background] Knieling F, Strobel D, Rompel O, Zapke M, Menendez-Castro C, Wolfel M, Schulz J, Rascher W, Jungert J. Spectrum, Applicability and Diagnostic Capacity of Contrast-Enhanced Ultrasound in Pediatric Patients and Young Adults after Intravenous Application - A Retrospective Trial. Ultraschall Med. 2016 Dec;37(6):619-626. doi: 10.1055/s-0042-108429. Epub 2016 Jun 14. PMID 27300274
- [Background] Stenzel M. Intravenous contrast-enhanced sonography in children and adolescents - a single center experience. J Ultrason. 2013 Jun;13(53):133-44. doi: 10.15557/JoU.2013.0014. Epub 2013 Jun 30. PMID 26674117
- [Background] Rafailidis V, Deganello A, Watson T, Sidhu PS, Sellars ME. Enhancing the role of paediatric ultrasound with microbubbles: a review of intravenous applications. Br J Radiol. 2017 Jan;90(1069):20160556. doi: 10.1259/bjr.20160556. Epub 2016 Sep 26. PMID 27610750